CLINICAL TRIAL: NCT04502901
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Healthy Male Subjects With Androgenetic Alopecia to Evaluate the Safety, Tolerability and PK of KX-826 Following Topical Multiple Dose Ascending
Brief Title: the Safety, Tolerability and PK of KX-826 in Healthy Males With Alopecia Following Topical Multiple Dose Ascending
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KX0826-US-1002
Record Dates: First submitted 2020-07-31; First posted 2020-08-06 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Group -KX0826 (Experimental): KX0826 is tropically applied to the scalp of healthy male subjects once a day for 14 days. The applied dosage cohorts are 2.5mg, 5mg, 10mg and 20mg.
  Interventions: Drug: KX0826
- Control Group- Placebo (Placebo Comparator): Placebo is tropically applied to the scalp of healthy male subjects once a day for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KX0826 — investigational AR antagonist
  Other Names: Pyrilutamide; KX-826
  Arms: Experimental Group -KX0826
Other: Placebo — Placebo of KX-826
  Arms: Control Group- Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability and PK of KX-826 following topical multiple ascending dose administration.

DETAILED DESCRIPTION:
KX-826 topical solution will be applied to the scalp of healthy male subjects with androgenetic alopecia.

A total of 40 subjects will be evaluated with 32 subjects randomized to receive active drug and 8 subjects randomized to receive placebo in a double-blind fashion (10 subjects in each dose cohort with 8 subjects randomized to receive active drug and 2 subjects randomized to receive placebo for a total of 4 dose cohorts).

Cohort Dose of KX-826 Subjects

1. 2.5 mg QD for 14 days 10 (8 active + 2 placebo)
2. 5 mg QD for 14 days 10 (8 active + 2 placebo)
3. 10 mg QD for 14 days 10 (8 active + 2 placebo)
4. 20 mg QD for 14 days 10 (8 active + 2 placebo)

Dose escalation will not occur until review of the multiple dose safety from the previous dose cohort is completed. Safety assessments will include monitoring of AEs, vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12-lead ECGs, skin irritation assessments and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are males between the ages of 18 and 60 years, inclusive;
3. Have a clinical diagnosis of androgenetic alopecia;
4. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs (systolic blood pressure ≥90 and ≤150 mmHg, diastolic blood pressure ≥50 and ≤95 mmHg and pulse rate ≥45 and ≤100 bpm; one repeat allowed to confirm out of range values);
5. Have normal renal and hepatic function as determined by the screening laboratory results;
6. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
7. Body mass index (BMI) of 19.0 to 35.0 kg/m2 inclusive and body weight not less than 50 kg;
8. Willing and able to adhere to study restrictions and to be confined at the CRU

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
2. Any visible skin disease, damage or condition at the application site which, in the opinion of the investigator, could compromise subject safety and/or interfere with the evaluation of the test site reaction;
3. Subject has any dermatological disorders of the scalp;
4. Subject has a history of hair transplants, hair weaves;
5. Subject has hypersensitivity to previously prescribed minoxidil or finasteride;
6. Known or suspected malignancy;
7. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody;
8. A hospital admission or major surgery within 30 days prior to screening;
9. Participation in any other investigational drug trial within 30 days prior to screening;
10. A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
11. A history of alcohol abuse according to medical history within 6 months prior to screening;
12. A positive screen for alcohol or drugs of abuse;
13. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
14. Use of prescription or over-the-counter (OTC) medications, and herbal (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at <3g/day is permitted until 24 hours prior to dosing);
15. An unwillingness of male participants to use appropriate contraceptive measures if engaging in sexual intercourse with a female partner of childbearing potential. Appropriate measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone subdermal implants, or a tubal ligation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) by skin irritation assessment, vital sign, ECG and clinical lab assessments | 19 days
  skin irritation assessment will be performed during the treatment period. The dermal response score will be based on a visual irritation scale (0-7) that rates the degree of erythema, edema and other signs of cutaneous irritation. abnormal vital sign (including blood pressure, pulse rate, respiratory rate and oral temperatures), 12-lead ECG, hematology (hemoglobin, hematocrit, platelet count, RBC count, WBC count, with differential), blood chemistry (BUN, creatinine, total bilirubin, alkaline phosphatase, AST, ALT, GGT, LDH, glucose, albumin, total protein, bicarbonate, phosphate, sodium, potassium, chloride, calcium, total cholesterol, uric acid) and urinalysis (pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrites, leukocytes, urobilinogen, microscopic urine analysis on abnormal findings) during the treatment period will be recorded and reported.
Incidence of study drug related TEAEs | 19 days
  incidence of study drug related TEAEs (possibly, probably or definitely)

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | 1 day
  Pharmacokinetics
Time at which Cmax was first observed (Tmax) | 1 day
  Pharmacokinetics
Area under the concentration curve from time 0 hour to 24 hour (AUC0-24) | 1 day
  Pharmacokinetics
Area under the concentration curve for on dosing interval at steady state (AUC0-t) | 19 days
  Pharmacokinetics
Cmax at steady state (Cmax_ss) | 19 days
  Pharmacokinetics
Time at which Cmax_ss was first observed (Tmax_ss) | 19 days
  Pharmacokinetics
Minimum observed or "trough" concentration at steady state (Cmin_ss) | 19 days
  Pharmacokinetics
Average concentration at steady state (Cav_ss) | 19 days
  Pharmacokinetics
AUC from time 0 and extrapolated to infinite time, total exposure (AUCinf) | 19 days
  Pharmacokinetics
AUC from time 0 to the last non-zero concentration (AUClast) | 19 days
  Pharmacokinetics
Biological half-life (T1/2 el) | 19 days
  Pharmacokinetics
Terminal elimination rate constant (Kel) | 19 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe Zhang, Study Director — Suzhou Kintor Pharmaceuticals Inc.
Locations (1):
- inVentiv Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No